CLINICAL TRIAL: NCT04223141
Title: Single-stapled Double Purse-string Anastomotic (SIA) Technique in Robotic Malignant Sigmoid Resections
Brief Title: Single-stapled Double Purse-string Technique for Colorectal Anastomosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIA2020
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Colo-rectal Cancer
Keywords: Robot
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): Robot-assisted laparoscopic resection of sigmoid colon with colorectal anastomosis constructed by the double purse-string technique
  Interventions: Procedure: SIA

INTERVENTIONS:
Procedure: SIA — As indicated by arm description

SUMMARY:
A single-arm, single-center prospective study of a novel double purse-string technique for constructing the colorectal anastomosis in robot-assisted laparoscopic resection of the sigmoid colon for cancer.

DETAILED DESCRIPTION:
In all, 30 consecutive patients will be enrolled. The first 5 will be regarded as a pilot series for testing and aligning the study setup. The next 25 patients will form the study group. The clinical outcomes will be compared with historical control patients from our own department. Safety and feasibility will be assessed by short-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria (all must be fulfilled):

* Verified cancer of the sigmoid colon
* Planned elective robot-assisted laparoscopic resection of sigmoid colon with primary anastomosis
* Operation with curative intent

Exclusion Criteria:

* Not legally competent and/or < 18 years old
* Not able to comprehend information and/or give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success | 30 days
  Successful construction of anastomosis by double purse-string technique
Complications | 30 days
  Surgical complications graded by Clavien-Dindo
Mortality | 30 days
  Postoperative death

SECONDARY OUTCOMES:
LOS | 90 days
  Length of stay - number of days from day of operation to discharge
Readmissions | 30 days
  Unplanned hospital admissions at least 24 hs after discharge
Operation time | 30 days
  Duration of operation from incision to last skin stitch
Blood loss | 30 days
  Estimated intraoperative blood loss in ml
Medical complications | 30 days
  Medical complications graded by Clavien-Dindo and MESS

CONTACTS AND LOCATIONS:
Overall Officials: Helene J Würtz, MD, Principal Investigator — Staff Surgeon; Flemming H Dall, MD PhD, Principal Investigator — Consultant; Hans B Rahr, MD DMSc, Study Director — Department Head
Locations (1):
- Vejle Hospital, Department of Surgery, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No